CLINICAL TRIAL: NCT00339989
Title: A Study to Understand Cervical Cancer Early Endpoints and Determinants (SUCCEED)
Brief Title: Cervical Cancer Early Endpoints and Determinants
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903302; 03-C-N302; NCT00558389 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cervical Cancer; Cervical Intraepithelial; Neoplasia; CIN
Keywords: Molecular Markers; Human Papillomavirus; Cervix; Cancer; Microarray
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Women undergoing colposcopy: women attending the University of Oklahoma Colposcopy Clinic

SUMMARY:
This study, conducted by the National Cancer Institute and the University of Oklahoma, will look for changes in cervix cells and other samples that may be signs of cervical disease. Human papilloma virus, or HPV, is a common infection of the genitalia in women that usually goes away by itself. If HPV infection does not go away, it might turn into cancer of the cervix, although this is rare. This study will examine why many HPV infections go away and why a few persist and lead to cervical cancer.

Women 18 years of age and older who are referred for colposcopy (examination of the vagina and cervix using an instrument with a magnifying lens) at the University of Oklahoma following Pap smear diagnosis may be eligible for this study. Women will be in one of the following diagnostic categories:

* Cancer: Stage 1-2 only.
* Precancer: Cervical intraepithelial neoplasia (CIN3).
* HPV-infected: Positive for any of the 13 known cancer-causing HPV types, but not diagnosed with cancer or CIN3.
* Normal: Negative for cancer-causing HPV and normal tissue laboratory results.

Participants will undergo the following procedures:

* Questionnaire: Covers demographic information (such as age, race, ethnicity, marital status, etc.), pregnancy history, menstrual and sexual history, contraceptive history, hormone medication history, medical history, smoking history, physical development, family history, and health care access.
* Blood test: 2 tablespoons of blood drawn.
* Colposcopy.
* Procedure to collect a sample of cervical cells and fluids for HPV testing and research.

DETAILED DESCRIPTION:
For the past twenty years, large epidemiologic natural history studies have played a crucial role in achieving our current understanding of cervical neoplasia. We now know that human papillomavirus (HPV) infection is necessary but not sufficient cause of cervical cancer. Cervical pathogenesis evolves as follows: normal 'yields' oncogenic HPV infection 'yields' precancer 'yields' invasive cancer. The majority of women with oncogenic HPV infections will not develop cancer, and most HPV infections, even those with associated cellular changes, regress in 1-2 years, probably eradicated or controlled by cellular immune response. Morevoer, while invasive cancer and precancer are histologically welldefined, the histological classification of low-grade lesions, now better defined as HPV infection, is very heterogeneous and poorly reproducible. Identifying women at highest risk for cancer prior to neoplastic progression is therefore a challenge. At present, we are unable to predict with any accuracy which HPV infections will progress and which are among the majority that regress. Currently, cytologic, histologic, and to some extent, HPV DNA assays are the basis for triage, treatment, and follow-up. While this approach has permitted successful cervical cancer prevention efforts, millions of women are diagnosed each year with HPV infections, and because of the inability to distinguish those who will progress from those who will regress, many women are over-treated as a result. It is therefore of etiologic interest and of public health benefit to develop a method for identifying the HPV-infected women at risk for progressing to precancer and invasion. To develop an accurate and reproducible division of precursor lesions (HPV infection and precancer) will require gaining knowledge about the molecular distinctions at each progressive disease state. Our goal is to therefore comprehensively assess biomarkers of risk for progressive cervical neoplasia, and thus develop a new set of biomarkers that can distinguish those at highest risk of cervical cancer from those with benign infection. Specifically, we will initially implement a cross-sectional study to develop a comprehensive list of potential risk biomarkers by examining cervical tissues of women with normal, HPV infection, precancer, and cancer. They will measure gene expression profiles to gain an accurate and comprehensive in vivo picture of cervical neoplasia carcinogenesis. We propose to then validate the most promising identified candidate biomarkers in a prospective design by assessing their predictive values for key outcomes related to progression (HPV persistence, diagnosis of precancer) or non-progression (HPV clearance).

ELIGIBILITY:
* INCLUSION CRITERIA:

All women who are referred for cervical colposcopy to the University of Oklahoma will be considered eligible for the study. These women will be categorized into four groups: (i) cancer, (ii) precancer, (iii) HPV-infected, and (iv) normal. Cancers will be limited to women diagnosed with early cancer (Stage 1-2) to minimize potential disease effects. Precancers will be defined as women diagnosed histologically with cervical intraepithelial neoplasia 3 (CIN3). This is a highly specific and well-reproduced diagnosis which effectively represents carcinoma in situ. All women testing DNA positive for any of the 13 known oncogenic HPV types (HPV-infected), but not diagnosed with CIN3 or cancer (all stages) will be placed in the HPV-positive group. This group will therefore encompass all HPV-infected women diagnosed with either cervical intraepithelial neoplasia 1 (CIN1), CIN2, low grade squamous intraepithelial lesion (LSIL), atypical squamous cells of undetermined significance (ASCUS), atypical glandular cells of underdetermined significance (AGUS), or found cytologically normal. Women referred to the colposcopy clinic but found to be negative for oncogenic HPV and normal upon histological diagnoses will be eligible as normal controls; this approach will be an ethical method for collecting biopsies from essentially "normal" women as there are many benign "look alike" conditions that are ruled out in colposcopy clinics. While this group may not be a random sample of the general population, the use of specimens from these women as controls will ensure a group of women who are truly confirmed as having no neoplasia.

EXCLUSION CRITERIA:

Women attending the clinic solely for vaginal colposcopies will be excluded from the study. Women who are under 18 years of age or pregnant at the visit will also be excluded from the study. In addition, women who have had prior treatment (women coming to the clinic for a follow-up visit subsequent to treatment (women coming to the clinic for a follow-up visit subsequent to treatment or women coming for their initial clinic visit following pretreatment with chemotherapy or radiation) will be excluded. All women with known HIV or AIDS will be excluded from the study. This information will not be readily available unless the woman has previously been seen at the University of Oklahoma clinic. This event is considered rare; recent studies of HIV and AIDS by the University of Oklahoma from the same population have been terminated due to the lack of HIV/AIDS detected in the population.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolled women attending the University of Oklahoma Colposcopy Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 3013 (Actual)
Dates: Start 2003-09-12 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Histology from biopsy or surgery | Cross-sectional
  Cervical precancer and cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Bustin SA. Absolute quantification of mRNA using real-time reverse transcription polymerase chain reaction assays. J Mol Endocrinol. 2000 Oct;25(2):169-93. doi: 10.1677/jme.0.0250169. PMID 11013345
- [Background] Hildesheim A, Herrero R, Castle PE, Wacholder S, Bratti MC, Sherman ME, Lorincz AT, Burk RD, Morales J, Rodriguez AC, Helgesen K, Alfaro M, Hutchinson M, Balmaceda I, Greenberg M, Schiffman M. HPV co-factors related to the development of cervical cancer: results from a population-based study in Costa Rica. Br J Cancer. 2001 May 4;84(9):1219-26. doi: 10.1054/bjoc.2001.1779. PMID 11336474
- [Background] Liaw KL, Glass AG, Manos MM, Greer CE, Scott DR, Sherman M, Burk RD, Kurman RJ, Wacholder S, Rush BB, Cadell DM, Lawler P, Tabor D, Schiffman M. Detection of human papillomavirus DNA in cytologically normal women and subsequent cervical squamous intraepithelial lesions. J Natl Cancer Inst. 1999 Jun 2;91(11):954-60. doi: 10.1093/jnci/91.11.954. PMID 10359548
- [Derived] Wentzensen N, Walker J, Smith K, Gold MA, Zuna R, Massad LS, Liu A, Silver MI, Dunn ST, Schiffman M. A prospective study of risk-based colposcopy demonstrates improved detection of cervical precancers. Am J Obstet Gynecol. 2018 Jun;218(6):604.e1-604.e8. doi: 10.1016/j.ajog.2018.02.009. Epub 2018 Feb 17. PMID 29462629
- [Derived] Liu AH, Walker J, Gage JC, Gold MA, Zuna R, Dunn ST, Schiffman M, Wentzensen N. Diagnosis of Cervical Precancers by Endocervical Curettage at Colposcopy of Women With Abnormal Cervical Cytology. Obstet Gynecol. 2017 Dec;130(6):1218-1225. doi: 10.1097/AOG.0000000000002330. PMID 29112672